CLINICAL TRIAL: NCT06411925
Title: A Multi-center, Randomized, Double-blinded, Active-controlled, Non-inferiority, Phase 4 Trial to Evaluate the Efficacy and Safety of Atock Dry Syrup Sama With Acute Bronchitis Patients
Brief Title: The Efficacy and Safety of Atock Dry Syrup With Acute Bronchitis Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: SamA Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SA21901-2
Record Dates: First submitted 2024-05-02; First posted 2024-05-13 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Acute Bronchitis
MeSH Terms: conditions — Bronchitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atock Dry Syrup (Experimental)
  Interventions: Drug: Atock Dry Syrup with placebo patch
- tulobuterol patch (Active Comparator)
  Interventions: Drug: Tulobuterol patch with placebo dry syrup

INTERVENTIONS:
Drug: Atock Dry Syrup with placebo patch — Atock Dry syrup (TID) with placebo patch (QD)
  Arms: Atock Dry Syrup
Drug: Tulobuterol patch with placebo dry syrup — Tulobuterol patch (QD) with placebo dry syrup (TID)
  Arms: tulobuterol patch

SUMMARY:
Clinical Study to Evaluate the Efficacy and Safety of Atock Dry Syrup with Acute bronchial Patients

ELIGIBILITY:
Inclusion Criteria:

1. Children aged ≥6 months to <12 years old
2. Total Bronchitis Severity Scale excluding sputum(BSSEs) ≥4
3. Wheezing score ≥2
4. Subjects who present symptoms of Acute Bronchitis within 48 hours from screening visit
5. Subject with negative results in HbsAg or HCV Ab test within 6 months from screening visit

Exclusion Criteria:

1. Subjects with chronic respiratory diseases (e.g., asthma, COPD) or severe respiratory diseases (e.g., pneumonia, cystic fibrosis, influenza, active tuberculosis)
2. Subjects under treatment with corticosteroids, antibiotics medications
3. Subjects with severe hepatic and renal impairment
4. Subjects with a history of drug abuse
5. Subject with positive results in HIV Ab test

Ages: 6 Months to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 296 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
The rate of subjects whose symptoms improved based on the wheezing score at 3 days | 3 days treatment period
  The rating was: 0=No wheezing (None); 1=mild (End expiration with stethoscope); 2=moderate (Inspiration and expiration with stethoscope) and 3=severe (Audible without stethoscope).

SECONDARY OUTCOMES:
The rate of subjects whose symptoms improved based on the wheezing score at 7 days | 7 days treatment period
The rate of subjects whose wheezing score improved by two or more grades at 3 and 7 days | 3 and 7 days treatment period
The change in bronchitis severity score excluding the sputum (BSSEs) at 3 and 7 days | 3 and 7 days treatment period
  • The BSSEs comprises the following four symptoms typical for Acute Bronchitis: cough, chest pain on coughing, crackle and dyspnea. These symptoms are each assessed according to a 5-point Likert scale: 0 = absent, 1 = mild, 2 = moderate, 3 = severe and 4 = very severe
The change in patient satisfaction scores for wheezing (VAS, Visual Analogue Scale) at 3 and 7 days | 3 and 7 days treatment period
  VAS consists of a horizontal line, usually 100 in length and select a point on the scale indicating the level of satisfaction for wheezing in the 3 and 7 days. The number 0 indicates not satisfaction and 100 indicates very satisfaction.
The change in patient satisfaction scores for cough (COAT, COugh Assessment Test) at 3 and 7 days | 3 and 7 days treatment period
  All items can be scored as a single scale (0-4 scaling of each item, 0-20 total score range). Higher scores represent more severe cough.

CONTACTS AND LOCATIONS:
Locations (1):
- Soonchunhyang University Seoul Hospital, Seoul, South Korea